CLINICAL TRIAL: NCT03107208
Title: Management of Diabetic Ketoacidosis in Children: Does Early Glargine Prevent Rebound Hyperglycemia?
Brief Title: Early Glargine (Lantus) in DKA Management in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1965
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Ketoacidosis; Type 1 Diabetes Mellitus
Keywords: DKA; type 1 diabetes; children; continuous glucose monitoring
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early glargine (Lantus) (Experimental): A dose of glargine (Lantus®) is given subcutaneously early in the management of DKA (i.e. while the participant is still receiving intravenous insulin). Participants will also be asked to wear a continuous glucose monitor (CGM) during the DKA and for a week following the DKA.
  Interventions: Drug: Glargine; Device: Continuous Glucose Monitor (Abbott FreeStyle Libre Pro)
- Control group (Other): A dose of glargine (Lantus®) is given subcutaneously after resolution of the DKA (i.e. when the intravenous insulin is stopped). This is currently the standard-of-care practice for children in DKA. Participants will also be asked to wear a continuous glucose monitor (CGM) during the DKA and for a week following the DKA.
  Interventions: Drug: Glargine; Device: Continuous Glucose Monitor (Abbott FreeStyle Libre Pro)

INTERVENTIONS:
Drug: Glargine — A dose of glargine (Lantus) will be given subcutaneously either early in the management of DKA (study group) or upon resolution of DKA (control group).
  Other Names: Lantus
Device: Continuous Glucose Monitor (Abbott FreeStyle Libre Pro) — All participants will be asked to wear a continuous glucose monitor (CGM) during the DKA and for a week following the DKA in order to better understand blood glucose control during DKA. This is an optional part of the study.
  Other Names: CGM

SUMMARY:
A frequent complication in the management of diabetic ketoacidosis (DKA) in children with type 1 diabetes is rebound hyperglycemia (blood glucose over 180 mg/dL) which increases the risk of re-developing DKA and can lengthen the hospital stay. The investigators want to study whether giving the long-acting insulin glargine (Lantus®) early in DKA management (versus after complete resolution of the DKA) helps prevent rebound hyperglycemia and makes the transition to insulin injections easier. Participants will also have the option to wear a continuous glucose monitor (CGM) during the study to help us understand blood glucose control during and after DKA.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) remains the leading cause of morbidity and mortality in children with type 1 diabetes (T1D) and the incidence of T1D is increasing. A frequent complication in DKA management that is associated with in-hospital mortality and longer hospital stay is hyperglycemia; specifically rebound hyperglycemia (defined as a serum glucose greater than 180 mg/dL) within 12-24 hours after correction of the DKA. Rebound hyperglycemia increases the patient's risk of re-developing DKA. Few adult studies suggest that giving the long-acting insulin analog (glargine or Lantus®) early in the management of DKA (i.e. while still receiving intravenous insulin) can reduce rebound hyperglycemia without an increased risk of hypoglycemia and result in a smoother transition from intravenous insulin to subcutaneous insulin. This has not been well-studied in children to date. In this study the investigators want to determine whether giving glargine early in DKA management in children results in reduced rebound hyperglycemia without an increased risk in hypoglycemia. The investigators will do this by randomizing participants in DKA to either receive glargine early in the management of DKA (study group) or after resolution of DKA (control group); the latter is currently standard-of-care. Additionally, continuous glucose monitoring (CGM) systems have not been studied in a pediatric population with DKA. These devices measure blood sugar levels every 5 minutes and provide a great deal of information about blood sugar control patterns over many days. Not only will the use of CGM in this study provide meaningful information regarding blood sugar patterns during DKA treatment, it will also broaden the investigators knowledge of whether CGM is a feasible and accurate tool to use in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-17.9 years at time of enrollment.
2. Known history of type 1 diabetes or presumed new-onset type 1 diabetes.
3. Diagnosis of DKA (serum glucose or fingerstick glucose concentration ≥ 200 mg/dL.
4. Venous pH ≤7.3 and/or serum bicarbonate concentration ≤15 mmol/L.
5. Evidence of ketonemia or ketonuria).

Exclusion Criteria:

1. Participants who present in DKA with conditions that affect neurological function such as:

   1. suspected alcohol or drug use,
   2. severe head trauma,
   3. meningitis, etc., who would not be able to consent/assent for the study.
2. Participants who present in DKA who are showing signs of altered mental status at time of enrollment.
3. Other known complicating illness or poorly-controlled chronic illness that is known to affect blood glucose levels and/or electrolyte balance such as:

   1. chronic renal disease (requiring hemodialysis),
   2. chronic liver disease (with evidence of current hepatic dysfunction,
   3. coagulopathy, and/or chronic hepatitis), or
   4. severe chronic lung disease (requiring the use of oral steroids).
4. Use of medications that are known to affect blood glucose levels such as:

   1. oral glucocorticoids,
   2. Metformin,
   3. SGLT2 inhibitors,
   4. GLP-1 receptor agonists,
   5. DPP-4 inhibitors,
   6. thiazolidinediones
   7. sulfonylureas, and
   8. vasopressors, etc.
5. Participants who have begun DKA treatment prior to being approached for enrollment and have received more than 6 hours of IV insulin therapy.
6. Participants who are known to be pregnant.
7. Participants who have a known diagnosis of type 2 diabetes.
8. Participants for whom the treating physicians feel a specific insulin regimen is necessary such that patient safety or well-being could be compromised by enrollment into the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ohman-Hanson, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants screen failed after consent form was signed.
Period: Overall Study
Arm/Group | Early Glargine (Lantus) | Control Group
Started | 30 | 27
Received Intervention | 26 | 24
Completed | 26 | 24
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Glargine (Lantus) | Control Group | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.3 [10.0 to 14.6] | 12.0 [9.75 to 14.7] | 12 [10 to 14.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 27 | 23 | 50
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
Diabetic patient status [Count of Participants; unit: Participants] — Whether the patient was newly diagnosed with type 1 diabetes (first presentation) or had a known diagnosis of T1D.
  Participants
    Newly diagnosed T1D | 11 | 11 | 22
    Known diagnosis of T1D | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Rate of Rebound Hyperglycemia
Description: Evaluate the rate of rebound hyperglycemia with a glucometer, defined as a serum glucose level of greater than 180 mg/dL (>10 mmol/L) within 12 hours after discontinuation of IV insulin, in children treated for diabetic ketoacidosis (DKA) with early glargine versus standard-of-care management. The number of patients that met this threshold is reported.
Time Frame: Within 12 hours after discontinuation of IV insulin
Measure: Count of Participants; unit: Participants
Arm/Group | Early Glargine (Lantus) | Control Group
Number analyzed (Participants) | 26 | 24
Participants | 20 | 18

2. Secondary Outcome: Rate of Recurrent Ketogenesis
Description: Evaluate the rate of recurrent ketogenesis (beta-hydroxybutyrate ≥ 1.5 mmol/L within 12 hours after discontinuation of IV insulin) in children treated for diabetic ketoacidosis (DKA) with early glargine versus standard-of-care management. The number of patients that met this threshold is reported.
Time Frame: Within 12 hours after discontinuation of IV insulin
Measure: Count of Participants; unit: Participants
Arm/Group | Early Glargine (Lantus) | Control Group
Number analyzed (Participants) | 26 | 24
Participants | 4 | 1

3. Secondary Outcome: Risk of Hypoglycemia Between Those Given Early Administration of Glargine Versus Those Given Standard-of-care Management.
Description: Assessment of the frequency of hypoglycemic events during treatment of DKA, and within 12 hours after discontinuation of IV insulin, in children given early glargine versus standard-of-care management vs. the rate of blood glucose decrease while receiving IV insulin in children with DKA given early glargine versus standard-of-care management. The number of participants who experienced hypoglycemia is reported.
Time Frame: During treatment and within 12 hours after d/c IV insulin; while receiving IV insulin in children with DKA given early glargine versus standard-of-care management.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Glargine (Lantus) | Control Group
Number analyzed (Participants) | 26 | 24
Participants | 4 | 2

4. Secondary Outcome: Evaluation of CGM and POC Glucose Monitoring During DKA Treatment in Children.
Description: Evaluation of the feasibility of CGM as a tool to monitor blood glucose levels during DKA treatment in children. The number of participants who consented to wear and placed the CGM is reported.
Time Frame: During treatment of DKA and within 12 hours after discontinuation of IV insulin.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Glargine (Lantus) | Control Group
Number analyzed (Participants) | 26 | 24
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Description: Only participants who received the intervention were monitored for adverse events. Adverse events specific to whether the participant agreed to wear a CGM were not monitored or assessed.
Arm/Group | Early Glargine (Lantus) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 7/26 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Glargine (Lantus) (N=26) | Control Group (N=24)
Hypoglycemia (Endocrine disorders) | 4 (4) | 2 (2)
Hypokalemia (Endocrine disorders) | 1 (1) | 0 (0)
Recurrent Ketosis (Endocrine disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03107208/Prot_SAP_000.pdf